CLINICAL TRIAL: NCT04372290
Title: CSD190401: An In-Clinic Confinement Study to Assess Elements of Abuse Liability for Nicotine-containing Pouch Tobacco Products
Brief Title: CSD190401: A Study to Assess Elements of Abuse Liability for Nicotine-containing Pouch Tobacco Products
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RAI Services Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CSD190401
Record Dates: First submitted 2020-04-29; First posted 2020-05-04 (Actual); Last update posted 2020-09-25 (Actual); Status verified 2020-09

CONDITIONS: Smoking; Smoking Behaviors; Tobacco Use; Tobacco Smoking
MeSH Terms: conditions — Smoking; Tobacco Use; Tobacco Smoking | interventions — HTR3D protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- Product usage order ABECD (Experimental): Subjects will use each of the 5 products sequentially (ABECD) during an evaluation period, followed by a 6 hour Test Session.
  Interventions: Other: Product A; Other: Product B; Other: Product C; Other: Product D; Other: Product E
- Product usage order BCADE (Experimental): Subjects will use each of the 5 products sequentially (BCADE) during an evaluation period, followed by a 6 hour Test Session.
  Interventions: Other: Product A; Other: Product B; Other: Product C; Other: Product D; Other: Product E
- Product usage order CDBEA (Experimental): Subjects will use each of the 5 products sequentially (CDBEA) during an evaluation period, followed by a 6 hour Test Session.
  Interventions: Other: Product A; Other: Product B; Other: Product C; Other: Product D; Other: Product E
- Product usage order DECAB (Experimental): Subjects will use each of the 5 products sequentially (DECAB) during an evaluation period, followed by a 6 hour Test Session.
  Interventions: Other: Product A; Other: Product B; Other: Product C; Other: Product D; Other: Product E
- Product usage order EADBC (Experimental): Subjects will use each of the 5 products sequentially (EADBC) during an evaluation period, followed by a 6 hour Test Session.
  Interventions: Other: Product A; Other: Product B; Other: Product C; Other: Product D; Other: Product E
- Product usage order DCEBA (Experimental): Subjects will use each of the 5 products sequentially (DCEBA) during an evaluation period, followed by a 6 hour Test Session.
  Interventions: Other: Product A; Other: Product B; Other: Product C; Other: Product D; Other: Product E
- Product usage order EDACB (Experimental): Subjects will use each of the 5 products sequentially (EDACB) during an evaluation period, followed by a 6 hour Test Session.
  Interventions: Other: Product A; Other: Product B; Other: Product C; Other: Product D; Other: Product E
- Product usage order AEBDC (Experimental): Subjects will use each of the 5 products sequentially (AEBDC) during an evaluation period, followed by a 6 hour Test Session.
  Interventions: Other: Product A; Other: Product B; Other: Product C; Other: Product D; Other: Product E
- Product usage order BACED (Experimental): Subjects will use each of the 5 products sequentially (BACED) during an evaluation period, followed by a 6 hour Test Session.
  Interventions: Other: Product A; Other: Product B; Other: Product C; Other: Product D; Other: Product E
- Product usage order CBDAE (Experimental): Subjects will use each of the 5 products sequentially (CBDAE) during an evaluation period, followed by a 6 hour Test Session.
  Interventions: Other: Product A; Other: Product B; Other: Product C; Other: Product D; Other: Product E

INTERVENTIONS:
Other: Product A — Usual brand (UB) filtered, combustible cigarette
Other: Product B — Nicorette® White Ice Mint 2 mg nicotine gum
Other: Product C — CSD1904-01, a nicotine pouch, 2 mg nicotine
Other: Product D — CSD1904-02, a nicotine pouch, 4 mg nicotine
Other: Product E — CSD1904-02, a nicotine pouch, 8 mg nicotine (simultaneous use of two 4 mg nicotine pouches)

SUMMARY:
This is a single site, open-label, randomized, cross-over study designed to evaluate elements of abuse liability (AL) including subjective effects and physiological measures (pharmacodynamics [PD]) and plasma nicotine uptake (pharmacokinetics [PK]) during and following ad libitum use of the study investigational products (IPs) by generally healthy subjects.

DETAILED DESCRIPTION:
Cigarette smokers (SMK) and smokers who also use smokeless tobacco (SST) [e.g., snus, moist snuff] will be recruited into the study. An attempt will be made to have approximately one third of the study population made up of SST.

Potential subjects may complete a pre-Screening telephone interview and will complete a Screening Visit to assess their eligibility within 45 days prior to check-in and enrollment/randomization.

Starting on Day -1, eligible subjects will begin confinement at the clinical site for 6 days. Subjects will be randomized to evaluate one investigational product (IP) in each of five separate Test Sessions, such that each subject will evaluate five IPs, including three strengths of the nicotine pouches, and both a high- and a low-AL comparator.

Each Test Session will last for approximately 4 hours during and following IP use and will include collection of both PD measures (subjective and physiological) and PK measures.

On Day -1, subjects will participate in an IP acclimation period where they will be instructed on how to use the nicotine pouch IP and the nicotine gum (low-AL comparator IP). At the end of the acclimation period, subjects will have access to their usual brand (UB) cigarettes for ad libitum use until the 12-hour tobacco abstinence begins prior to the Day 1 Test Session.

ELIGIBILITY:
Inclusion Criteria:

1. Able to read, understand, and willing to sign an informed consent form (ICF) and complete questionnaires written in English.
2. Generally healthy male or female, 21 to 60 years of age, inclusive, at the time of consent.
3. Expired breath carbon monoxide level is ≥ 10 ppm and ≤ 100 ppm at Screening.
4. Positive urine cotinine test at Screening.
5. Smokes combustible, filtered, non-menthol or menthol cigarettes, 83 mm to 100 mm in length as primary source of tobacco. Other cigarette sizes may be allowed with sponsor approval.
6. Smokers who also use smokeless tobacco products may be enrolled.
7. Agrees to smoke same UB cigarette throughout the study period. UB cigarette is defined as the reported cigarette brand style currently smoked most frequently by the subject.
8. Smokes at least 10 cigarettes per day (on average) and inhales the smoke, for at least 6 months prior to Screening.
9. Response at Screening to Fagerström Test for Nicotine Dependence (FTND) Question 1 ("How soon after you wake up do you smoke your first cigarette?") is either "Within 5 minutes" or "6-30 minutes."
10. Willing to use UB cigarette, nicotine pouch products, and Nicorette gum during the study period.
11. Willing to abstain from tobacco and nicotine use for at least 12 hours prior to each Test Session.
12. Females must be willing to use a form of contraception acceptable to the Principal Investigator (PI) from the time of signing informed consent until End-of-Study.
13. Agrees to in-clinic confinement of 6 days (5 nights).

Exclusion Criteria:

1. Uses a vapor product (e.g., e-cigarettes, tank systems) more than one day per week, for the past 6 months prior to screening.
2. Presence of clinically significant uncontrolled cardiovascular, pulmonary, renal, hepatic, endocrine, gastrointestinal, psychiatric, hematological, neurological disease, or any other concurrent disease or medical condition that, in the opinion of the PI, makes the study subject unsuitable to participate in this clinical study.
3. History, presence of, or clinical laboratory test results indicating diabetes.
4. Systolic blood pressure of > 160 mmHg or a diastolic blood pressure of > 95 mmHg, measured after being seated for five minutes at Screening and at Day -1.
5. Weight of ≤ 110 pounds.
6. Hemoglobin level is < 12.5 g/dL for females or <13.0 g/dL for males at Screening.
7. Scheduled treatment for asthma currently or within the past consecutive 12 months prior to the Screening Visit. As-needed treatment, such as inhalers, may be included at the PI's discretion pending approval from the Medical Monitor.
8. Positive test for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C virus (HCV).
9. Any history of cancer, except for primary cancers of skin such as localized basal cell/squamous cell carcinoma that has been surgically and/or cryogenically removed.
10. Use of any medication or substance that aids in smoking cessation, including but not limited to any nicotine-replacement therapy (NRT) (e.g., nicotine gum, lozenge, patch), varenicline (Chantix®), bupropion (Wellbutrin®, Zyban®), or lobelia extract within (≤) 30 days prior to the signing of informed consent.
11. History or presence of bleeding or clotting disorders.
12. Any use of anticoagulants or aspirin (≥ 325 mg/day).
13. Whole blood donation within 8 weeks (≤ 56 days) prior to the signing of informed consent.
14. Plasma donation within (≤) 7 days prior to the signing of informed consent.
15. Participation in another clinical trial within (≤) 30 days prior to the signing of informed consent. The 30-day window for each subject will be derived from the date of the last study event in the previous study to the time of signing the informed consent form (ICF) in the current study.
16. Females who have a positive pregnancy test, are pregnant, breastfeeding, or intend to become pregnant during the course of the study.
17. Individuals ≥ 35 years of age currently using systemic, estrogen-containing contraception or hormone replacement therapy.
18. A positive urine drug screen without evidence of prescribed corresponding concomitant medication(s) at Screening or Day -1.
19. Postpones a decision to quit using tobacco- or nicotine-containing products in order to participate in this study or a previous attempt within (≤) 30 days prior to signing the ICF.
20. Drinks more than 21 servings of alcoholic beverages per week or has a positive alcohol screen result at Screening or Day -1.
21. Employed by a tobacco or nicotine company, the study site, or handles tobacco- or nicotine-containing products as part of their job.
22. Determined by the PI to be inappropriate for this study.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2020-05-06 (Actual); Primary Completion 2020-06-04 (Actual); Study Completion 2020-06-04 (Actual)

PRIMARY OUTCOMES:
AUECPL 5-240 | 5 minutes to 240 minutes
  area-under-the-effects curve (AUEC) for PL numeric rating scale (NRS) score-versus-time curve from 5 minutes to 240 minutes after the start of IP use.
Emax PL | 240 minutes
  maximum product liking (PL) numeric rating scale (NRS) score after the start of IP use.

CONTACTS AND LOCATIONS:
Overall Officials: Bobbette Jones, DrPH, Study Director — RAIS
Locations (1):
- New Orleans Center for Clinical Research (NOCCR), Knoxville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No